CLINICAL TRIAL: NCT06860672
Title: Safety, Tolerability and Preliminary Efficacy Study of a Single Intrathecal Injection of the Dual Vector AAV-CHD3-R1025W Base Editor for the Treatment of Developmental Disorders Caused by the R1025W Mutation in the CHD3 Gene
Brief Title: Clinical Trial of the Dual Vector Base Editor for the Treatment of the CHD3-R1025W Mutation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yongguo Yu (Other)
Responsible Party: Sponsor-Investigator, Yongguo Yu, Chief physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-25-002
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Developmental Delay Disorder; Intellectual Disability; Rare Diseases
MeSH Terms: conditions — Developmental Disabilities; Intellectual Disability; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dual vector treatment group (Experimental)
  Interventions: Genetic: Dual vector DNA base editor

INTERVENTIONS:
Genetic: Dual vector DNA base editor — The base editor is delivered using a dual vector adeno-associated virus (AAV) system and introduced into the child via intrathecal injection to correct the mutated CHD3 gene. The vital signs of the child will be closely monitored during treatment to assess possible acute adverse effects. The child will be followed up regularly after treatment to monitor the success of gene editing and the neurodevelopmental improvement of the child. Possible long-term adverse events will be closely monitored to assess the safety of the treatment.

SUMMARY:
To evaluate the safety, tolerability and preliminary efficacy study of a single intrathecal injection of the dual vector AAV-CHD3-R1025W base editor for the treatment of developmental disorders caused by the R1025W mutation in the CHD3 gene

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Snijders Blok-Campeau syndrome
* Heterozygous mutation of c.3073C>T, p.(Arg1025Trp) in the CHD3 gene
* Normal liver, heart and immune function
* Normal coagulation and platelet counts

Exclusion Criteria:

* Brain tumor or intracranial space-occupying lesion
* Contraindications to administration of lumbar puncture or sheath injection administration
* Persistent status epilepticus or recurrent epileptic control instability
* Presence of unstable systemic disease including active bacterial, fungal or HIV, hepatitis A, hepatitis B infection
* Serum anti-AAV neutralizing antibody titer >1:50 (ELISA immunoassay)
* Treatment with immunological agents other than protocol-specified prophylaxis within 3 months
* Prior gene therapy
* Participation in another clinical trial, or treatment with another investigational product within 30 days or 5 half-lives
* Known allergy to any investigational product

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of drug-related serious adverse events | 0-26 weeks

SECONDARY OUTCOMES:
Evaluate the changes using the Clinical Global impression Scale -Overall improvement (CGI-I) | 0-26 weeks
  This 7-point scale (1 = very much improved, 7 = very much worse, etc.) is used by the clinician to assess the participant's overall performance status; higher scores indicate increased severity.
Evaluate the changes in the Patient's Global Impressions of Improvement (PGI-I) scale | 0-26 weeks
  This 7-point scale (1 = very much improved, 7 = very much worse, etc.) is used by the clinician to assess the participant's overall performance status; higher scores indicate increased severity.

CONTACTS AND LOCATIONS:
Overall Officials: Yongguo Yu, Dr, MD, PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Zilong Qiu, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine Songjiang Research Institute
Locations (1):
- Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No